CLINICAL TRIAL: NCT04150770
Title: A Clinical Trial of Infliximab for Injection in Refractory Childhood Uveitis
Brief Title: A Clinical Trial of Infliximab for Childhood Uveitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiaomin Zhang (Other)
Responsible Party: Sponsor-Investigator, Xiaomin Zhang, Principal Investigator, MD, PhD, Tianjin Medical University
Organization: Tianjin Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017KY-05
Record Dates: First submitted 2019-09-22; First posted 2019-11-05 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Uveitis; Infliximab
MeSH Terms: conditions — Uveitis | interventions — Infliximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | US Export: Yes

ARMS (1):
- Patients with Childhood Uveitis (Experimental): 5mg/kg/dose of infliximab IV initially two weeks, then 4 weeks and then every 6-8 weeks
  Interventions: Drug: infliximab

INTERVENTIONS:
Drug: infliximab
  Other Names: Remicade

SUMMARY:
This project is designed to test the hypothesis that infliximab is clinically useful for patients with refractory childhood uveitis.

DETAILED DESCRIPTION:
Approval of the study was obtained from the hospital's ethical committee. The study design and methodology followed the tenets of Declaration of Helsinki. All patients were provided with written informed consent and received a thorough explanation of the study design, aims, and the off-label use of infliximab, its potential risks and benefits. This is a prospective non-comparative interventional study.

Participants will receive intravitreal injections of suggested dose of infliximab (5 mg/kg/dose) and data will be collected prospectively with regard to ophthalmologic outcomes. Study participants will be followed for up to 10 months to determine efficacy and side effects, and an additional 30 days for safety reports. Descriptive statistics will be gathered on participant demographics, uveitis characteristics, change in immunosuppressive medications, number of responders, ophthalmologic measures and change in corticosteroid dose during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Ages 4 to 18 years old,
* Non-infectious uveitis
* Persistent uveitis uncontrolled by topical medications, or unacceptable side effects of topical medications.
* Failure of at least six weeks of treatment with a non-biological disease modifying agent such as methotrexate, cyclosporine, mycophenolate mofetil, or azathioprine.
* Ability to provide informed consent (subject or parent/guardian)
* Onset of uveitis < 16 years of age.
* Topical ophthalmologic treatments allowed.
* Systemic corticosteroid use at entry may be allowed.
* Participant must be able to cooperate for a non-sedated slit lamp exam and visual acuity examination.
* Negative Purified Protein Derivative (PPD) placed and read within 1 month of initiation of infliximab
* The screening laboratory test results must meet the following criteria:

WBC (white blood cell count): within normal range for institution ANC (absolute neutrophil count): within normal range for institution Hemoglobin: greater than 10 grams/deciliter Platelets: within normal range for institution Serum Creatinine: within normal range for age AST - aspartate aminotransferase - within normal range for institution ALT - alanine aminotransferase- within normal range for institution

Exclusion Criteria:

* Previous use of biologic medications for uveitis.
* Intraocular steroid injection or ophthalmologic surgery within the preceding 3 months.
* Uveitis due to trauma or intraocular surgery
* A history of a known allergy to murine products.
* Documentation of seropositivity for human immunodeficiency virus (HIV).
* Documentation of a positive test for hepatitis B surface antigen or hepatitis C
* A known history of a serious infection (e.g., hepatitis, pneumonia, or pyelonephritis) in the previous 3 months.
* An opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening.
* A concomitant diagnosis or history of congestive heart failure.
* A history of lymphoproliferative disease.
* Any known malignancy or a history of malignancy.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.
* Use of any investigational drug within 30 days prior to screening or within five half-lives of the first dose of the investigational agent, whichever is longer.
* Presence of a transplanted solid organ.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change In LogMAR Best Corrected Visual Acuity (BCVA) From Baseline to Each Visit. | 24 weeks
  Participant's best corrected visual acuity was measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR chart. On the logMAR scale, 0 is equivalent to 20/20 visual acuity, the range of normal vision is considered to be from -0.2 - 0.1; higher values indicate visual impairment.

SECONDARY OUTCOMES:
Change in Anterior Chamber (AC) Cell Grade From Baseline to Each Visit. | 24 weeks
  Slit lamp examinations were conducted at each visit to assess AC cell count. The number of AC cells observed within a 1 mm × 1 mm slit beam was used to determine the grade according to the Standardization of Uveitis Nomenclature (SUN) criteria:
  Grade 0 = < 1 cell Grade 0.5+ = 1 - 5 cells Grade 1+ = 6 - 15 cells Grade 2+ = 16 - 25 cells Grade 3+ = 26 - 50 cells Grade 4+ = > 50 cells.
Change in Vitreous Haze (VH) Grade From Baseline to Each Visit. | 24 weeks
  Vitreous haze was measured using dilated indirect ophthalmoscopy (DIO) and assessed by the Investigator according to National Eye Institute (NEI) and SUN criteria:
  Grade 0: No evident vitreous haze; Grade 0.5+: Slight blurring of the optic disc margin because of the haze; normal striations and reflex of the nerve fiber layer cannot be visualized; Grade 1+: Permits a better definition of both the optic nerve head and the retinal vessels (compared to higher grades); Grade 2+: Permits better visualization of the retinal vessels (compared to higher grades); Grade 3+: Permits the observer to see the optic nerve head, but the borders are quite blurry; Grade 4+: Optic nerve head is obscured.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomin Zhang, M.D., Study Director — Tianjin Medical University Eye Hospital

IPD SHARING:
Plan to Share IPD: No
Study protocol, statistical analysis plan and informed Consent form can be shared with other researchers.